CLINICAL TRIAL: NCT05531240
Title: Transurethral Prostate Resection (TURP) vs. Prostate Artery Embolization (PAE): Open Multicentric Randomized Study for Evaluation of Outcomes, Complications, and Health Economics
Brief Title: Transurethral Prostate Resection (TURP) vs. Prostate Artery Embolization (PAE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Centrallasarettet Västerås (Other); Lasarettet i Enköping (Other); Sormland County Council, Sweden (Other); Helsingborgs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 276725
Record Dates: First submitted 2022-05-30; First posted 2022-09-07 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Transurethral Resection of Prostate Syndrome; Prostate Hyperplasia; Embolization, Therapeutic
Keywords: Prostate embolisation; PAE
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAE (Experimental): Prostate Artery Embolization (PAE)
  Interventions: Procedure: Prostate Artery Embolization
- TURP (Active Comparator): Transurethral Prostate Resection (TURP)
  Interventions: Procedure: Transurethral Prostate Resection (TURP)

INTERVENTIONS:
Procedure: Prostate Artery Embolization — Prostate Artery Embolization (PAE) is performed by experienced interventional radiologists. The method involves catheterization of the prostate vessels superselectively with two to three French microcatheters. PAE is performed with microspheres of 250 to 400 µm in size.
  Arms: PAE
Procedure: Transurethral Prostate Resection (TURP) — Under general/regional anesthesia, a resectoscope is inserted into the urethra that carries an electric metal loop (monopolar or bipolar diathermy) that is used to cut and extract the prostate tissue.
  Arms: TURP

SUMMARY:
This study focuses on the treatment of benign prostatic hyperplasia which causes lower urinary tract symptoms.

The purpose of the research project is to evaluate PAE in terms of both medical and health economic outcomes. To evaluate whether there are any differences in effect (IPSS), complications, costs and perceived quality of life compared with TUR-P.

ELIGIBILITY:
Inclusion Criteria:

* Benign prostatic hyperplasia where medical treatment has not helped or for other reasons has not been deemed applicable
* IPSS>=8
* Prostate volume [40-80] ml measured via transrectal ultrasound
* Peak flow rate (Qmax) <= 15 ml / s,
* Verified obstruction by urodynamic studies (cystometry)
* Surgery not contraindicated

Exclusion Criteria:

* Prostate cancer
* Severe atherosclerosis
* Kidney failure
* Urethral stricture
* Active cystitis or prostatitis
* Bladder stone.
* Neurogenic bladder disorder
* Contrast product allergy

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of lower urinary tract symptoms | 24 months
  Assess the change in the lower urinary tract symptoms using the International Prostate Symptom Score (IPSS) questionnaire before and after prostate artery embolization procedure (PAE) compared to transurethral resection of the prostate (TURP)
Health care costs | 24 months
  Assess the health care costs after prostate artery embolization procedure (PAE) compared to transurethral resection of the prostate (TURP)

SECONDARY OUTCOMES:
Adverse effects, | 24 months
  Assess the adverse effects after prostate artery embolization procedure (PAE) compared to transurethral resection of the prostate (TURP)
Quality of life (Short Form Health Survey [EQ-5D-5L ]) | 24 months
  Assess the quality of life after prostate artery embolization procedure (PAE) compared to transurethral resection of the prostate (TURP). Scored 0-100, where 0 is the lowest and 100 the highest possible quality of life.
Erectile function | 24 months
  Erectile function using the International Index of Erectile Function (IIEF-5). The possible scores for the IIEF-5 range from 5 to 25, and ED is classified into five categories based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25).
Prostate-Specific Antigen (PSA) | 24 months
  Assess the change in PSA

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Chabok, Principal Investigator — CKF Västerås Uppsala university
Locations (4):
- Sweden (4):
  - Helsingborgs Hospital, Helsingborg, Region Skånes
  - Mälarsjukhuset, Eskilstuna, Region Sörmland
  - Lasarettet i Enköping, Enköping, Region Uppsala
  - Region Vastmanland Hospital, Västerås, Västmanland County

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Garraway WM, Collins GN, Lee RJ. High prevalence of benign prostatic hypertrophy in the community. Lancet. 1991 Aug 24;338(8765):469-71. doi: 10.1016/0140-6736(91)90543-x. PMID 1714529
- [Background] Hunter DJ, McKee M, Black NA, Sanderson CF. Health status and quality of life of British men with lower urinary tract symptoms: results from the SF-36. Urology. 1995 Jun;45(6):962-71. doi: 10.1016/s0090-4295(99)80116-2. PMID 7539561
- [Background] Barry MJ, Fowler FJ Jr, O'Leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT. The American Urological Association symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Association. J Urol. 1992 Nov;148(5):1549-57; discussion 1564. doi: 10.1016/s0022-5347(17)36966-5. PMID 1279218
- [Background] Young S, Golzarian J. Prostate embolization: patient selection, clinical management and results. CVIR Endovasc. 2019 Jan 18;2(1):7. doi: 10.1186/s42155-019-0049-1. PMID 32027007
- [Background] Burnett AL, Wein AJ. Benign prostatic hyperplasia in primary care: what you need to know. J Urol. 2006 Mar;175(3 Pt 2):S19-24. doi: 10.1016/S0022-5347(05)00310-1. PMID 16458735
- [Background] Pinheiro LC, Martins Pisco J. Treatment of benign prostatic hyperplasia. Tech Vasc Interv Radiol. 2012 Dec;15(4):256-60. doi: 10.1053/j.tvir.2012.09.004. PMID 23244720
- [Background] Carnevale FC, Antunes AA, da Motta Leal Filho JM, de Oliveira Cerri LM, Baroni RH, Marcelino AS, Freire GC, Moreira AM, Srougi M, Cerri GG. Prostatic artery embolization as a primary treatment for benign prostatic hyperplasia: preliminary results in two patients. Cardiovasc Intervent Radiol. 2010 Apr;33(2):355-61. doi: 10.1007/s00270-009-9727-z. Epub 2009 Nov 12. PMID 19908092
- [Background] McWilliams JP, Bilhim TA, Carnevale FC, Bhatia S, Isaacson AJ, Bagla S, Sapoval MR, Golzarian J, Salem R, McClure TD, Kava BR, Spies JB, Sabharwal T, McCafferty I, Tam AL. Society of Interventional Radiology Multisociety Consensus Position Statement on Prostatic Artery Embolization for Treatment of Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia: From the Society of Interventional Radiology, the Cardiovascular and Interventional Radiological Society of Europe, Societe Francaise de Radiologie, and the British Society of Interventional Radiology: Endorsed by the Asia Pacific Society of Cardiovascular and Interventional Radiology, Canadian Association for Interventional Radiology, Chinese College of Interventionalists, Interventional Radiology Society of Australasia, Japanese Society of Interventional Radiology, and Korean Society of Interventional Radiology. J Vasc Interv Radiol. 2019 May;30(5):627-637.e1. doi: 10.1016/j.jvir.2019.02.013. Epub 2019 Mar 27. No abstract available. PMID 30926185
- [Background] Gao YA, Huang Y, Zhang R, Yang YD, Zhang Q, Hou M, Wang Y. Benign prostatic hyperplasia: prostatic arterial embolization versus transurethral resection of the prostate--a prospective, randomized, and controlled clinical trial. Radiology. 2014 Mar;270(3):920-8. doi: 10.1148/radiol.13122803. Epub 2013 Nov 13. PMID 24475799
- [Background] Abt D, Hechelhammer L, Mullhaupt G, Markart S, Gusewell S, Kessler TM, Schmid HP, Engeler DS, Mordasini L. Comparison of prostatic artery embolisation (PAE) versus transurethral resection of the prostate (TURP) for benign prostatic hyperplasia: randomised, open label, non-inferiority trial. BMJ. 2018 Jun 19;361:k2338. doi: 10.1136/bmj.k2338. PMID 29921613
- [Background] NICE Guidance - Prostate artery embolisation for lower urinary tract symptoms caused by benign prostatic hyperplasia: (c) NICE (2018) Prostate artery embolisation for lower urinary tract symptoms caused by benign prostatic hyperplasia. BJU Int. 2018 Jul;122(1):11-12. doi: 10.1111/bju.14404. No abstract available. PMID 29894572
- See also: Guidelines on Management of Non-Neurogenic Male Lower Urinary Tract Symptoms (LUTS), incl. Benign Prostatic Obstruction (BPO) 2021. I: European Association of Urology Guidelines 2021 Edition — https://uroweb.org/guideline/treatment-of-non-neurogenic-male-luts